CLINICAL TRIAL: NCT06273514
Title: TECAR Therapy Might be an Alternative to Dry Needling in the Treatment of Active Myofascial Trigger Points in Upper Trapezius
Brief Title: Comparison the Effects of TECAR With Dry Needling in the Treatment of Myofascial Trigger Points
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Silesia (Other)
Responsible Party: Principal Investigator, Tomasz Piętka, School of Health Sciences in Katowice, Department of Physical Medicine, Chair of Physiotherapy, Medical University of Silesia in Katowice, Poland, Medical University of Silesia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TECAR and DN intervention
Record Dates: First submitted 2024-02-07; First posted 2024-02-22 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Myofascial Pain Syndrome of Neck; Myofascial Trigger Point Syndrome; Myofascial Trigger Point Pain
Keywords: myofascial trigger point; myofascial pain syndrome; TECAR therapy; dry needling; upper trapezius.
MeSH Terms: conditions — Fibromyalgia; Myofascial Pain Syndromes | interventions — Dry Needling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TECAR (Experimental): TECAR therapy is a non-invasive method for treating musculoskeletal system disorders based on the application of high-frequency current (300 kHz - 1 MHz)
  Interventions: Other: TECAR
- Dry needling (Experimental): Dry needling, a form of intramuscular stimulation, is a therapeutic intervention employed in physiotherapy and sports medicine. It entails the precise insertion of fine needles into specific myofascial trigger points, taut bands of skeletal muscle, or connective tissue without the administration of pharmacological agents.
  Interventions: Other: Dry needling

INTERVENTIONS:
Other: TECAR — TECAR therapy performs using a WINBACK® 1s device (Daeyang Medical Co. Ltd, South Korea) with a maximum power of 100W. A 500 kHz frequency capacitive electrode is applied directly to the active MTrP in the UT. The closed electrode is placed distally on the arm. Lowpulse modulation use during treatment with half-second pauses. This enables the application of the current directly into the MTrP without enrolling the entire muscle. The single exposure last for 10 min. The current dose participant-dependent and ranged from 40 to 60% (100% = 100 Watts).
  Each time, before and after treatment, and 30 days after the first therapy, the following features will be asses: pain intensity, muscle strength, and ROM.
  Other Names: capacitive and resistive transfer of energy
  Arms: TECAR
Other: Dry needling — Dry needling performs using SOMA needles (25 mm x 0.3 mm). During the therapy, the participant is in a prone position. The affected UT region is disinfect before needling. The taut band localizes between the thumb and index finger of the researcher. The needle within the plastic guide tube is place over the MTrP at the UT. The needle directly inserts into the MTrP. A local twitch response confirms the accuracy of the puncture. Needling performs using Hong's "fast in, fast out" technique. The needle will be withdrawn if no twitching will observe.
  Other Names: DN
  Arms: Dry needling

SUMMARY:
The aim of the study is to assess the effectiveness of dry needling (DN) and capacitive and resistive transfer of energy (TECAR) therapy in the treatment of myofascial trigger points (MTrPs) as well comparison of their efficacy.

Research hypothesis:

Capacitive and resistive energy transfer therapy is comparable to dry needling therapy for the treatment of myofascial trigger points.

It is estimated that the presence of trigger points is the main cause of pain in 30-85% of patients visiting primary health care facilities and pain management clinics. The presence of trigger points may significantly affect the patient's functional status and daily functioning. Recently, diagnostic criteria and methods of treating trigger points have evolved significantly. However, the usefulness of different imaging methods in the diagnosis of trigger points has not yet been established. Despite numerous studies, the long-term effectiveness of the dry needling method is still unknown. Furthermore, there is no available research on the short- and long-term effectiveness of capacitive and resistive energy transfer therapy in the treatment of trigger points.

Therefore, the objectives of the work were:

Determination and comparison of the short- and long-term effects of capacitive and resistive energy transfer therapy and the dry needling technique of myofascial trigger points located in the upper trapezius muscle (UT) on the strength, neck range of motion and pain intensity within this muscle.

The study is planned to include a group of 26 men aged 25 to 45 who suffer from pain caused by the presence of myofascial trigger points in the upper trapezius muscle. The subjects will be divided into two groups of equal number of people. The first group will undergo therapy using the dry needling technique, while the second group will undergo capacitive and resistive energy transfer therapy.

In order to determine the immediate effects of capacitive and resistive energy transfer therapy and dry needling techniques, measurements of muscle strength, the intensity of pain in the upper trapezius muscle and neck range of motion will be performed before and after each therapeutic session (2 session in 2 weeks are planed). In turn, to determine the long-term effects of capacitive and resistive energy transfer therapy and dry needling, the next above-mentioned measurements will be performed four weeks after the end of first therapy.

ELIGIBILITY:
Inclusion Criteria:

* sex male
* age 25-45
* manually confirmed active MTrP in the upper trapezius

Exclusion Criteria:

* MTrP therapy in the upper trapezius region during the last year
* history of neck trauma
* history of cervical spine surgeries
* history of humeral joint surgeries
* cervical radiculopathy
* chronic and acute diseases of the cardiovascular system
* chronic and acute diseases of the respiratory system
* chronic and acute diseases of the nervous systems
* endocrine disturbances
* skin lesions in upper trapezius area
* acute inflammation
* cancer
* BMI > 30 kg/m2.

Ages: 25 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Pain - Pressure pain threshold (PPT) | The measurements were performed three times with a 30-second break. The results are presented as the mean value of these measurements and are expressed in kg/m2.
  Defined as the minimum force applied which induces pain, asses using an algometer BioFEET V3 (MusTec, Almere, Netherlands). The head of the algometer was placed on the MTrP in the upper trapezius (UT) and then pressed until the participant verbally expressed their PPT.
Pain - numerical rating scale (NRS) | Up to 3 minutes before and up to 3 minutes after each interventions
  This pain screening tool uses a 0-10 scale, with 0 indicating no pain and 10 indicating the worst imaginable pain.

SECONDARY OUTCOMES:
Muscle strength | Measurements will be perform three times on both sides of the body up to 5 minutes before and up to 5 minutes after each interventions . The highest results obtained for statistical analysis and will be expressed as kG (kilogram force)
  Measures using a dynamometer (BioFEET V3; -MusTec, Muscle Dynamic Technology BV, Louis Chrispijnstraat1, Netherlands 1325 PC ALMERE). We assume that scapula elevation is the indicatory movement for the UT. During the assessment, the humeral joint remained in a natural position with proximal stabilization. The head of the dynamometer will be then placed on the acromion. The physiotherapist resisted active movements to provoke isometric contraction of the UT.
Cervical spine range of motion (ROM) | Each movement will be perform three times up to 10 minutes before and up to 10 minutes after each interventions. The results are present as the mean value of these measurements and are express in degrees (°)
  Cervical spine ROM was measured using a goniometer (BASEline). The following movements were assessed: flexion, extension, rotation, and side bending.
  During the measurements the participants sit. While measuring cervical spine flexion and extension, the axis of the goniometer is place on the auricle opening. During the rotation, the axis of the goniometer is place at the top of the skull. Side bends measures with the goniometer axis placed on the spinal process of the axis (C2).

CONTACTS AND LOCATIONS:
Locations (1):
- Medical fit, Ruda Śląska, Silesian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No